CLINICAL TRIAL: NCT06671769
Title: Natural Heart Health Supplement Trial
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 34661
Record Dates: First submitted 2024-10-28; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Cholesterol; Cholesterol (total and HDL)
Keywords: heart health

STUDY DESIGN:
Intervention Model Description: The "Natural Heart Health Supplement Trial" is designed as a single-arm treatment study, where participants will serve as their own controls. This innovative approach, termed a "Signal Phase" study at Efforia, aims to evaluate the potential efficacy and safety of an experimental natural heart health supplement over a 3-month period. Participants will consume a daily dose of the supplement, which is administered in a chocolate-flavored powdered format. The primary objective is to assess the impact of the supplement on key heart health biomarkers, including Total Cholesterol, HDL-C, LDL-C, Triglycerides, and High-Sensitivity C-reactive protein (hs-CRP). By utilizing this methodology, the study will provide preliminary insights into the supplement's effects, offering a directional indication of potential positive results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Natural Heart Health Dietary Supplement in Chocolate Powder Form (Experimental): a natural heart-health dietary supplement in chocolate powder form designed to be taken daily.
  Interventions: Dietary Supplement: Heart Health Supplement

INTERVENTIONS:
Dietary Supplement: Heart Health Supplement — This is a natural heart health supplement in powdered format, chocolate flavor where participants will take a daily dose.

SUMMARY:
We are running a 3-month trial of an experimental natural heart health supplement. Participants will take a daily dose of an experimental natural heart health supplement in powdered format, chocolate flavor. The trial will assess changes in heart biomarkers such as Total Cholesterol, HDL-C, LDL-C, Triglycerides, and High-Sensitivity C-reactive protein (hs-CRP).

DETAILED DESCRIPTION:
Heart disease is a leading cause of death in the United States, and maintaining healthy cholesterol levels is crucial for heart health. While social media and the press have focused on trendier treatments for general longevity, for most of us keeping our cholesterol in check will make a major impact. Research indicates that natural substances long used in Eastern medicine, can positively affect cholesterol levels and reduce inflammation, both vital for cardiovascular wellness.

This study aims to empower participants with evidence-based insights about the effectiveness of a natural heart health supplement in managing cholesterol levels and reducing inflammation. By participating, you'll contribute to valuable research while potentially enhancing your heart health through natural means.

This study aims to assess the impact of a natural heart health supplement on Total Cholesterol, HDL-C, LDL-C, Triglycerides, and hs-CRP levels over three months. Our objective is to provide evidence supporting or refuting the supplement's efficacy.

ELIGIBILITY:
Exclusion Criteria:

* Individuals with known soy allergies
* Individuals with liver disease
* Pregnant or breastfeeding individuals

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Total Cholesterol | from Baseline to 30 day and 90 day.
  Total Cholesterol as measured by an at-home blood collection kit returned to the lab
HDL Cholesterol | from baseline to 30 day and 90 day
  as measured by an at-home blood collection kit returned to the lab
LDL Cholesterol | Baseline to 30 day and 90 day
  as measured by an at-home blood collection kit returned to the lab
Triglycerides | From baseline to 30 day and 90 day
  as measured by at-home blood collection returned to lab

SECONDARY OUTCOMES:
hs-CRP | from baseline to 30 day and 90 day
  as measured by at-home blood test returned to a lab.

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia - Study will be entirely online, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided